CLINICAL TRIAL: NCT02640092
Title: Longitudinal Evaluation of [18F]GTP1 as a PET Radioligand for Imaging Tau in the Brain of Patients With Prodromal, Mild, and Moderate Alzheimer's Disease Compared to Healthy Volunteers
Brief Title: Longitudinal Evaluation of [18F]GTP1 as a PET Radioligand for Imaging Tau in the Brain of Participants With Alzheimer's Disease Compared to Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GN30009; G0097 (Other: InVicro)
Record Dates: First submitted 2015-12-15; First posted 2015-12-28 (Estimated); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — (18F)GTP1

ARMS (1):
- [18F]GTP1 (Experimental): Participants will complete [18F]GTP1 PET imaging at four time points: Baseline, 6 months, 12 months and 18 months. For each [18F]GTP1 imaging session, the following procedure will be performed: a catheter will be placed for intravenous (IV) administration of [18F]GTP1. Participants will receive an IV bolus injection of up to 370 megabecquerel (MBq) (10 millicurie [mCi]) of [18F]GTP1.
  Interventions: Drug: [18F]GTP1

INTERVENTIONS:
Drug: [18F]GTP1 — Participants will receive [18F]GTP1 as per the schedule specified in the arm description.
  Other Names: [18F]G02941054; [18F]MNI-798; [18F]RO6880276

SUMMARY:
This is an open-label, longitudinal observational study evaluating the imaging characteristics of the tau positron-emission tomography (PET) radioligand [18F] Genentech Tau Probe 1 (GTP1) in the brain of participants with prodromal, mild, and moderate Alzheimer's disease (AD) compared to healthy participants. The overall goal of this protocol is to evaluate the longitudinal change in tau burden using [18F]GTP1, a tau targeted radiopharmaceutical.

ELIGIBILITY:
Inclusion Criteria:

For All Participants:

- Availability of a study partner who, in the investigator's judgment, has frequent and sufficient contact with the participant and is able to provide accurate information regarding the participant's cognitive and functional abilities, agrees to accompany the participant and provide information at visits

For Healthy Participants:

* Healthy with no clinically relevant finding on physical examination at screening and upon reporting for the Baseline [18F]GTP1 imaging visit
* Have no cognitive complaint
* Have a Clinical Dementia Rating Scale (CDR) global score = 0
* Have a Mini-Mental State Examination (MMSE) score of 28-30

For Participants With a Diagnosis of AD:

* Participants with mild or moderate AD must meet National Institute on Aging - Alzheimer's Association (NIA-AA) core clinical criteria for probable AD dementia, with an amnestic presentation
* Participants with prodromal AD must meet NIA-AA core clinical criteria for mild cognitive impairment (MCI)
* Have screening [18F]florbetapir PET imaging demonstrating amyloid binding based on qualitative visual read
* A brain MRI consistent with a diagnosis of AD, with no evidence of non-AD disease to account for dementia or MRI exclusion criteria
* Medications taken for symptomatic treatment of AD must remain stable for at least 30 days prior to screening visit
* Satisfy one of the following subgroups: Approximately 20 prodromal AD (MMSE 24-30, CDR = 0.5); Approximately 20 mild AD (MMSE 22-30, CDR = 0.5 or 1); Approximately 20 moderate AD (MMSE 16-21, CDR = 0.5 or 1 or 2)

Exclusion Criteria:

* Current or prior history of any drug or alcohol abuse
* Participants with any significant psychiatric, neurological, or unstable medical disorder expected to interfere with the study
* Participants unable to undergo MRI and PET scan
* For participants contributing CSF samples, any contraindication to lumbar puncture
* Prior participation in other research protocols or clinical care in the last year such a radiation exposure combined with that from the present study exceeds an effective dose of 50 millisievert (mSV), the allowable annual limit for research participants as stipulated by the Food and Drug Administration (FDA)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-06-11 (Actual)

PRIMARY OUTCOMES:
Change in Standardized Uptake Value Ratio (SUVR) as Measured by [18F]GTP1 | From Baseline to 18 months

SECONDARY OUTCOMES:
Correlation Coefficient Between Change in SUVR (as Measured by [18F]GTP1) and Change in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog)13 | From Baseline to 18 months
Correlation Coefficient Between Change in SUVR (as Measured by [18F]GTP1) and Change in Volumetric Magnetic Resonance Imaging (MRI) Measures | From Baseline to 18 months
Correlation Coefficient Between Change in SUVR (as Measured by [18F]GTP1) and Change in Cerebrospinal Fluid (CSF) Markers | From Baseline to 18 months
Percentage of Participants With Adverse Events (AEs) | From Baseline to 18 months
Test-Retest Variability Based on [18F]GTP1 PET Scans | From date of test scan to 7-21 days after test scan

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- United States (16):
  - Molecular NeuroImaging, New Haven, Connecticut
  - KI Health Partners, LLC; New England Institute for Clinical Research, Stamford, Connecticut
  - Neuropsychiatric Research; Center of Southwest Florida, Fort Myers, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - Bioclinica Research, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - NeuroStudies.net, LLC, Decatur, Georgia
  - Acadia Clinical Research; Dr. Henderson's Office, Bangor, Maine
  - Donald S. Marks, M.D., P.C.; Medical Center, Plymouth, Massachusetts
  - Alzheimers Disease Center, Quincy, Massachusetts
  - NeuroCognitive Institute, Mount Arlington, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Advanced Medical Research, Maumee, Ohio
  - Lehigh Center Clinical Research, Allentown, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Sanabria Bohorquez SM, Baker S, Manser PT, Tonietto M, Galli C, Wildsmith KR, Zou Y, Kerchner GA, Weimer R, Teng E. Evaluation of partial volume correction and analysis of longitudinal [18F]GTP1 tau PET imaging in Alzheimer's disease using linear mixed-effects models. Front Neuroimaging. 2024 Mar 28;3:1355402. doi: 10.3389/fnimg.2024.1355402. eCollection 2024. PMID 38606196
- [Derived] Teng E, Manser PT, Sanabria Bohorquez S, Wildsmith KR, Pickthorn K, Baker SL, Ward M, Kerchner GA, Weimer RM. Baseline [18F]GTP1 tau PET imaging is associated with subsequent cognitive decline in Alzheimer's disease. Alzheimers Res Ther. 2021 Dec 1;13(1):196. doi: 10.1186/s13195-021-00937-x. PMID 34852837
- [Derived] Blennow K, Chen C, Cicognola C, Wildsmith KR, Manser PT, Bohorquez SMS, Zhang Z, Xie B, Peng J, Hansson O, Kvartsberg H, Portelius E, Zetterberg H, Lashley T, Brinkmalm G, Kerchner GA, Weimer RM, Ye K, Hoglund K. Cerebrospinal fluid tau fragment correlates with tau PET: a candidate biomarker for tangle pathology. Brain. 2020 Feb 1;143(2):650-660. doi: 10.1093/brain/awz346. PMID 31834365